CLINICAL TRIAL: NCT05755139
Title: Safety and Efficacy Evaluation of SMART Camera Treatment Presets for Cutaneous Lesions Using IPL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lumenis Be Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LUM-ABU-SMRT-22-01
Record Dates: First submitted 2022-11-29; First posted 2023-03-06 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-04

CONDITIONS: Vascular Lesion; Pigmented Lesions

STUDY DESIGN:
Intervention Model Description: Single Group Assignmen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- IPL with smart diagnostic handpiece (Experimental): Standard IPL module which has FDA clearance (K083733) for a wide range of indications including vascular and pigmented lesions. The Universal IPL handpiece (HP) operates at a spectrum of 400-1,200 nm with 7 different cut-off filters and 2 different notch filters that can be easily inserted into the handpiece to treat different conditions.
  The SMART Camera is a novel add-on skin diagnostic (SD) tool. The SD module includes a proprietary spectral camera embedded in a handpiece, and proprietary computer vision-based algorithms designed to process the spectral information and to determine the skin attributes and optimal treatment IPL preset.
  Interventions: Device: IPL with smart diagnostic handpiece

INTERVENTIONS:
Device: IPL with smart diagnostic handpiece — treatment with IPL following diagnostic with SMART system

SUMMARY:
Multi-center, Prospective, Open-Label with Before-After Study Design. Each subject will receive a single treatment. Treatment presets will be determined by the SMART Camera system and approved by the physician. Follow-up will take place at 1 month following the treatment. Skin and lesion attributes will be examined by the SMART system and the physician

DETAILED DESCRIPTION:
At least 40 healthy subjects in 2 sites, aged 21-80 years old with visible textural lesions including but not limited to Lentigines, Rosacea, and Age spots / Telangiectasia on the face or décolletage that wish to improve their skin appearance. Each patient should have at least 3 treatment areas (e.g. left cheek, right cheek, forehead, nose, chin, upper/lower décolletage) that contains at least one type of lesion

ELIGIBILITY:
Inclusion Criteria:

* 1. Healthy Female/Male, age 21-80. 2. Fitzpatrick skin type I-V. 3. Presence of visible textural lesions including but not limited to:

  * Lentigines
  * Rosacea (erythematotelangiectatic rosacea and papulopustular rosacea)
  * Age spots/Telangiectasia
  * Telangiectasia 4. Patients should have at least 3 treatment areas of the following: right cheek, left cheek, forehead, nose, chin, and upper/lower décolletage. 5. Able to read, understand and provide written Informed Consent. 6. Able and willing to comply with the treatment/follow-up schedule and requirements.

    7. Willing to have digital photographs taken of all of the treatment areas before, during, and after treatment. 8. Willing to refrain from using any prescription or over-the-counter topical creams used for the treatment of veins or pigmented lesions in the treatment area during the study period.

    9. Willing to protect and/or have very limited sun exposure and use an approved sunscreen of SPF 50 or higher in the treatment area, every day for the duration of the study. 10. Agree not to undergo any other procedure(s) in the same treatment areas during the study.

    11. Women of child-bearing age are required to be using a reliable method of birth control (such as an intrauterine device, birth control pills, condom with spermicidal, NuvaRing, partner with vasectomy, or abstinence) at least 3 months prior to enrollment and throughout the course of the study.

Exclusion Criteria:

* Any of the following will exclude the subject from the study:

  1. Previous treatments on the same area/s at least six months prior to screening
  2. Skin type VI
  3. Pregnant, intending to become pregnant during the course of study, less than 3 months postpartum or less than 6 weeks after completion of breastfeeding
  4. Exposure to the sun or artificial tanning during 3-4 weeks prior to treatment. Any remaining suntan, sunburn, or artificial tanning products.
  5. Active infections in the treatment area
  6. Dysplastic nevi
  7. Significant concurrent skin conditions or any inflammatory skin conditions
  8. Active cold sores, open lacerations, or abrasions
  9. Chronic or cutaneous viral, fungal or bacterial diseases
  10. Treatment should not be attempted on patients with a history or concurrent condition of skin cancer or pre-cancerous lesions in the treatment area
  11. Tattoos in the areas to be treated

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-12-04 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
To study the safety of the suggested treatment presets as suggested by the SMART IPL system platform for cutaneous lesions in subjects with skin types I-V | 3 month
  Treatment with the SMART IPL system will be considered safe when a full treatment is completed using the recommended presets by the AI system (presets are not overruled due to safety by the physician) with no serious AEs. The overall percentage of safe treatments using the AI-recommended presets from all treatments will be calculated through study completion, an average of 3 months.
To study the efficacy of the SMART IPL system for cutaneous lesions treatment in subjects with skin types I-V | 4 months
  Lesions clearance will be evaluated by the investigator at a 1-month follow-up compared to baseline using a 5-point clearance scale, when 0 is no clearance, and 4 is 76-100% clearance.
  Evaluation will be completed through study completion, an average of 4 months.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Friedmann, MD, Principal Investigator — Westlake dermatology; Jennifer Deaver, Principal Investigator — The Pearl Dermatology
Locations (2):
- United States (2):
  - Westlake Dermatology, Austin, Texas
  - The Pearl Dermatology, Houston, Texas